CLINICAL TRIAL: NCT06430294
Title: Force-time Characteristics of Spinal Mobilizations Delivered on Pediatric Manikins
Brief Title: Caracteristics of Pediatric Spinal Mobilizations
Status: Recruiting | Type: Observational
Sponsor: Université du Québec à Trois-Rivières (Other)
Responsible Party: Principal Investigator, Isabelle Pagé, Professor, Université du Québec à Trois-Rivières
Other Study IDs: UQTR_IP_SIMULATIONS_2024
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Spinal Mobilization
Keywords: Chiropractic; Pediatric; Simulations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Chiropractors will perform spinal mobilizations on three different pediatric-sized manikins while a sensor will measure the force and time parameters used.
  Interventions: Other: Spinal mobilisation

INTERVENTIONS:
Other: Spinal mobilisation — Application of a force on pediatric manikins.

SUMMARY:
This observational study aims to create simulations using pediatric manikins to teach pediatric spinal mobilizations. We'll measure the force and duration of spinal mobilizations applied by chiropractors on pediatric manikins. Another objective is to gather feedback from both students and teachers on the effectiveness of using manikins for teaching.

The main questions it aims to answer are:

1. How much force and for how long do chiropractors apply spinal mobilizations on pediatric manikins?

DETAILED DESCRIPTION:
This project aims to initiate the development of low-fidelity simulations to enhance the learning of skills associated with performing pediatric spinal mobilizations. This will be achieved by gathering target values for the force and duration of spinal mobilizations performed by chiropractors on pediatric manikins.

ELIGIBILITY:
Inclusion Criteria:

* Being a chiropractor in private practice and a member of the Ordre des chiropraticiens du Québec

Exclusion Criteria:

* Not been able to perform pediatric spinal mobilizations

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Licensed chiropractors
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Peak force (N) reached during the spinal mobilization measured by a force sensor | During the spinal mobilization
  The spinal mobilization will be delivered on a force sensor (Loadpad(R)) that will measured the force-time characteristics. The peak force reached during the therapy will be extracted.
Duration (s) of spinal mobilization measured by a force sensor | During the spinal mobilization
  The spinal mobilization will be delivered on a force sensor (Loadpad(R)) that will measured the force-time characteristics. The duration of the therapy will be extracted.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Pagé, DC, PhD, Principal Investigator — Université du Québec à Trois-Rivières
Locations (1):
- Université Québec à Trois-Rivières, Trois-Rivières, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No